CLINICAL TRIAL: NCT03512977
Title: Effect of the Sphenopalatine Ganglion Block for Post Spinal Headache Treatment: A Prospective Randomized Controlled Study
Brief Title: Is Sphenopalatine Ganglion Block Treatment Effective on Postspinal Headaches
Acronym: SPG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayse Zeynep Turan, Principle investigator, Derince Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DerinceTRH-03
Record Dates: First submitted 2018-04-12; First posted 2018-05-01 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Headache Disorders; Central Nervous System Diseases
Keywords: spinal anesthesia; sphenopalatine ganglion block; postspinal headache
MeSH Terms: conditions — Headache Disorders; Central Nervous System Diseases; Post-Dural Puncture Headache | interventions — Sphenopalatine Ganglion Block; Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sphenopalatine Ganglion Block Group (Experimental): patients will be performed transnasal sphenopalatine block and conservative treatment ( iv hydration, analgesic agents, caffeine or theophylline)
  Interventions: Procedure: sphenopalatine ganglion block; Drug: conservative treatment
- Standard Treatment Group (Active Comparator): patients will receive standard supportive treatment ( Conservative treatments are iv hydration, analgesic agents, caffeine or theophylline)
  Interventions: Drug: conservative treatment

INTERVENTIONS:
Procedure: sphenopalatine ganglion block — the intervention will be performed on sitting position. Lidocaine 2% viscous (0.5ml) will be apply on cotton swab sticks and one will be gently inserted into nostril, along the floor of the nose. Stick will be used to insert it as far as it goes with the intention to reach the nasopharyngeal wall (posterior wall of the nose). At that position the swab stick will be left undisturbed for 20 minutes.
  Arms: Sphenopalatine Ganglion Block Group
Drug: conservative treatment — Conservative treatments are iv hydration, analgesic agents, caffeine or theophylline

SUMMARY:
This study evaluates effect of sphenopalatine ganglion block in post dural puncture headache. Half of participants will receive standard supportive treatment and other half of patients will be performed sphenopalatine ganglion block.

DETAILED DESCRIPTION:
Spinal anesthesia is known subarachnoid block also commonly used regional anesthesia technic. Spinal anesthesia is frequently performed in obstetric patients undergoing cesarian section, which has several advantages including less deep vein thrombosis incidence, low opioid requirement, early mobilization and early lactation also has some complications too. Postdural headache is one of the most known complications of spinal anesthesia.

The etiology of the postspinal headache remains unclear. Severeness of the symptoms and amount of the cerebrospinal fluid leakage have been found positive correlating. The cerebrospinal fluid supports brain with it's mass effect. When a leakage of the fluid occurs, support of the brain decreases and pain sensitive structures of the brain gets more sensitive. In this condition 5 th 9th and 10 th cranial nerves, falks cerebelli, tentorium and blood vessels are affected most. Decreased cerebrospinal fluid volume causes decreased brain volume and compensatory mechanisms lead to cerebral venous dilatation. Conservative treatments are iv hydration, analgesic agents, caffeine or theophylline. Epidural blood patch is the gold standard for the treatment . However epidural blood patch is an invasive technic and has some complications such as dural puncture, infection and neurologic trauma.

Sphenopalatine ganglion is one of the four parasympathetic thin ganglion in skull. Parasympathetic fibers innervates cerebral and meningeal blood vessels which cause vasodilatation and stimulate nociceptor activation on meninges. Consequently headache is related with sensory cortex.

Transnasal SPG block is performed successfully in chronic pain syndromes including migraine, cluster headaches and atypic face pain. Likewise the SPG block is performed in acute treatment of postspinal headache. However gold standard of the treatment is epidural blood patching which is interventional and has many risks. Several studies enrolled limited participants offer SPG block primarily in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Patients who was diagnosed for postdural puncture headache after cesarian section
* Patients who is fluent speaking and writing in turkish

Exclusion Criteria:

* Refusal to participate in the study
* Patients who was known lidocaine sensitivity
* Patients with severe nasal septum deviation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale Score | 24 th hour after intervention
  VAS score will be asked to the patients. Visual analog scale (VAS) from 0 to 10. 0(= no anxiety), 10(= highest level of anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: mehmet yilmaz, Study Director — Sağlık Bilimleri Üniversitesi Kocaeli Derince Eğitim ve Araştırma Hastanesi
Locations (1):
- Derince Research and Training Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No